CLINICAL TRIAL: NCT04705337
Title: Levosimendan In Ambulatory Heart Failure Patients
Acronym: LEIA-HF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The level of recruitment, 62 participants enrolled, does not allow for achieving the protocol-defined target of 350 participants by the end of the recruitment period.
Sponsor: Medical University of Bialystok (Other)
Collaborators: Medical Research Agency, Poland (Other Government); University of Opole (Other); Medical University of Lodz (Other); Poznan University of Medical Sciences (Other); Nicolaus Copernicus University (Other); National Institute of Cardiology, Warsaw, Poland (Other); Azienda Ospedaliera dei Colli (Other); John Paul II Hospital, Krakow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/ABM/01/00017
Record Dates: First submitted 2021-01-04; First posted 2021-01-12 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure New York Heart Association Class III; Heart Failure New York Heart Association Class IV; Heart Failure, Systolic; Heart Failure With Reduced Ejection Fraction
MeSH Terms: conditions — Heart Failure, Systolic | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levosimendan (Experimental): administration of levosimendan
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator): administration of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levosimendan — administration of levosimendan as a continuous iv. infusion, every 4 weeks for 48 weeks (12 infusions in total)
  Arms: Levosimendan
Other: Placebo — administration of glucose as a continuous iv. infusion, every 4 weeks for 48 weeks (12 infusions in total)
  Arms: Placebo

SUMMARY:
The objective of the study is to determine the efficacy of repeated infusions of levosimendan in the group of outpatients with advanced systolic heart failure (HF).

DETAILED DESCRIPTION:
It is a multicentre, randomized, double-blind, placebo-controlled study. 350 subjects will be included (in 12 or more medical centers) with severe HF, ejection fraction ≤35%, in New York Heart Association class III or IV. The other inclusion criteria concern: hospitalization for the HF decompensation in the last 3 months and a reduced six-minute walk test <350m or elevated NTproBNP ≥1000 pg / mL. To the European Society of Cardiology-guided, individually optimized medical therapy (OMT) the investigational product (IP) will be added. The subjects will be randomly assigned to one of the study group: 175 to the levosimendan arm and 175 to the placebo arm. The intervention studied in LEIA-HF trial is the administration of levosimendan as a continuous iv. infusion, every 4 weeks for 48 weeks (12 infusions in total). All study participants will also continue OMT. In the second phase of the study, after completing the levosimendan / placebo infusions, another 6 visits are planned, still double-blind, every 4 weeks, to assess the safety of treatment discontinuation (with optional return to the infusions by the Investigator when additional criteria for HF decompensation are met).

The efficacy of the treatment will be assessed after 52 weeks, 4 weeks after the last levosimendan / placebo administration.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial activities
* Male or female, age ≥ 18 years at the time of signing informed consent
* Left ventricle ejection fraction ≤ 35%
* Hospitalization due to worsening of HF within the last 3 months
* New York Heart Association functional class III or outpatient IV
* Individually optimized pharmacotherapy, based on the current European Society of Cardiology recommendations, stable for at least 1 month prior to randomization, according to the knowledge and experience of the qualifying clinician
* Distance covered in six-minute walk test <350m OR NTproBNP concentration ≥ 1000 pg/mL
* In the opinion of the Investigator, the patient does not currently require hospitalization
* Patient protected with an implantable device capable of terminating life-threatening arrhythmias and conduction disturbances (ICD or cardiac resynchronisation therapy-D/P), if indicated and the patient consents to implantation.

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products,
* Restrictive or hypertrophic cardiomyopathy, uncorrected severe valvular disease, potentially reversible cause of HF
* Hypotension with symptoms of tissue hypoperfusion
* Uncontrolled hypertension
* Planned revascularization or other surgical treatment of HF within the next year
* Advanced chronic kidney disease
* Features of liver damage
* Severe chronic lung disease with features of respiratory distress or severe abnormal spirometry or home oxygen treatment
* Accompanying chronic diseases with poor prognosis
* Paroxysmal supraventricular tachycardia, paroxysmal ventricular tachycardia, torsade de pointes, advanced atrioventricular blocks within one month prior to screening
* Receipt of any investigational product within 30 days before screening visit
* Any disorder, which in the investigator's opinion may jeopardise subject's safety or compliance with the study protocol and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
the number of unplanned hospitalization | 12 months of follow-up period
  unplanned hospitalization due to heart failure decompensation
the number of deaths | 12 months of follow-up period
  death for any cause

SECONDARY OUTCOMES:
total mortality calculations | 0-12, 12-18 and 0-18 months
  total mortality for any cause
cardiovascular mortality calculations | 0-12, 12-18 and 0-18 months
  mortality due to cardiovascular reasons
the number of planned hospitalization | 0-12, 12-18 and 0-18 months
  planned hospitalization due to heart failure decompensation
the number of implantations of mechanical circulatory support | 0-12, 12-18 and 0-18 months
  implantation of mechanical circulatory support
the number of heart transplantations | 0-12, 12-18 and 0-18 months
  heart transplantation
quality of life measurements | 0-12, 12-18 and 0-18 months
  The Kansas City Cardiomyopathy Questionnaire quality of life questionnaire- an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
the six-minute walk test | 0-12, 12-18 and 0-18 months
  measures the distance an individual is able to walk over a total of six minutes
NTproBNP measurements | 0-12, 12-18 and 0-18 months
  measurements of NTproBNP concentrations
estimated glomerular filtration rate measurements | 0-12, 12-18 and 0-18 months
  measurements of estimated glomerular filtration rate
echocardiographic parameters | 0-12, 12-18 and 0-18 months
  the change in numerous echocardiographic parameters with different units assessed in each patient in transthoracic echocardiographic examination (TTE)
patients who returned to levosimendan / placebo infusions | from the 12th to the 18th months of the study
  calculations of the percentage of patients who returned to levosimendan / placebo infusions

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Tycińska, Prof. MD, Study Chair — Medical University of Bialystok; Marek Gierlotka, Prof. MD, Principal Investigator — University of Opole; Jarosław Kasprzak, Prof. MD, Principal Investigator — Medical University of Łódź; Jacek Kubica, Prof. MD, Principal Investigator — Nicolaus Copernicus University in Toruń; Grzegorz Grześk, Prof. MD, Principal Investigator — Nicolaus Copernicus University in Toruń; Jadwiga Nessler, Prof. MD, Principal Investigator — John Paul II Hospital, Krakow; Janina Stępińska, Prof. MD, Principal Investigator — Cardinal Stefan Wyszyński Institute of Cardiology; Ewa Straburzyńska-Migaj, Prof. MD, Principal Investigator — Poznan University of Medical Sciences
Locations (14):
- Poland (14):
  - Medical University of Bialystok Clinical Hospital, Bialystok
  - Medical University Hospital No.1, Bydgoszcz
  - Medical University Hospital No.2, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Górnośląskie Centrum Medyczne Śląskiego Uniwersytetu Medycznego, Katowice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - John Paul II Hospital, Krakow
  - Provincial Specialist Hospital named after Dr. Wł. Biegański, Lodz
  - Medical University Hospital, Opole
  - University Hospital of Lord's Transfiguration, Poznan
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Warsaw
  - Cardinal Stefan Wyszyński Institute of Cardiology, Warsaw
  - Uniwersytecki Szpital Kliniczny, Wroclaw
  - Śląskie Centrum Chorób Serca, Zabrze

IPD SHARING:
Plan to Share IPD: No
According to the agreement with the funding institution (Medical Research Agency), the sponsor and research centers must obtain the consent of the funding institution to disclose the clinical trial data.